CLINICAL TRIAL: NCT01288573
Title: A Phase 1/2 Combined Dose Ranging and Randomized, Open-label, Comparative Study of the Efficacy and Safety of Plerixafor in Addition to Standard Regimens for Mobilization of Haematopoietic Stem Cells Into Peripheral Blood, and Subsequent Collection by Apheresis, Versus Standard Mobilization Regimens Alone in Pediatric Patients, Aged 1 to <18 Years, With Solid Tumours Eligible for Autologous Transplants.
Brief Title: A Combined Study in Pediatric Cancer Patients for Dose Ranging and Efficacy/Safety of Plerixafor Plus Standard Regimens for Mobilization Versus Standard Regimens Alone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFI12860; 2010-019340-40 (EudraCT Number); MOZ15609 (Other: Genzyme other study code)
Record Dates: First submitted 2011-01-28; First posted 2011-02-02 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Ewing's Sarcoma/Soft Tissue Sarcoma; Neuroblastoma; Brain Tumors
MeSH Terms: conditions — Neuroblastoma; Brain Neoplasms | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Plerixafor 160 μg/kg (Experimental): Patients will receive subcutaneous (SC) injection of 160 μg/kg plerixafor in addition to their standard mobilization regimen. Each dose of plerixafor will be administered in the evening 9 to 11 hours prior to apheresis (up to a maximum of 5 apheresis sessions).
  Interventions: Drug: plerixafor
- Plerixafor 240 μg/kg (Experimental): Patients will receive subcutaneous (SC) injection of 240 μg/kg plerixafor in addition to their standard mobilization regimen. Each dose of plerixafor will be administered in the evening 9 to 11 hours prior to apheresis (up to a maximum of 5 apheresis sessions).
  Interventions: Drug: plerixafor
- Plerixafor 320 μg/kg (Experimental): Patients will receive subcutaneous (SC) injection of 320 μg/kg plerixafor in addition to their standard mobilization regimen. Each dose of plerixafor will be administered in the evening 9 to 11 hours prior to apheresis (up to a maximum of 5 apheresis sessions).
  Interventions: Drug: plerixafor

INTERVENTIONS:
Drug: plerixafor — 160 μg/kg subcutaneous (SC) injection
  Arms: Plerixafor 160 μg/kg
Drug: plerixafor — 240 μg/kg subcutaneous (SC) injection
  Arms: Plerixafor 240 μg/kg
Drug: plerixafor — 320 μg/kg subcutaneous (SC) injection
  Arms: Plerixafor 320 μg/kg

SUMMARY:
This is a multi-site study with plerixafor in pediatric cancer patients. The study will be conducted in 2 stages:

* Stage 1 is a dose-escalation study.
* Stage 2 is an open-label, randomized, comparative study using the appropriate dosing regimen identified in the Stage 1 dose-escalation study.

All participating patients will receive a standard mobilization regimen as per study site practice guidelines (either chemotherapy plus once daily granulocyte-colony stimulating factor (G-CSF) or once daily G-CSF alone). The only change to the standard mobilization regimen is the addition of plerixafor treatment prior to apheresis for all patients in Stage 1 (dose escalation), and for those patients randomized to the plerixafor plus standard mobilization treatment arm in Stage 2 (randomized, comparative).

Stage 1 will enroll at least 27 patients. Stage 2 will enroll at least 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to < 18 years during stage 1 and 1 to < 18 years during stage 2
* Ewing's sarcoma, soft tissue sarcoma, lymphoma, neuroblastoma, brain tumors or other malignancy (excluding any form of leukemia) requiring treatment with high dose chemotherapy and autologous transplant as rescue therapy
* Eligible for autologous transplantation
* Recovered from all acute significant toxic effects of prior chemotherapy
* Adequate performance status (for patients ≥16 years of age, defined as Karnofsky score >60 and for patients <16 years of age, defined as Lansky score >60)
* Absolute neutrophil count >0.75 × 10^9/L
* Platelet count >50 × 10^9/L
* Calculated creatinine clearance (using the Schwartz method): during study Stage 1, >80 mL/min/1.73m^2 and during study Stage 2, >60 mL/min/1.73m^2
* Aspartate aminotransferase(AST)/serum glutamic oxaloacetic transaminase(SGOT), alanine aminotransferase(ALT)/serum glutamic pyruvic transaminase (SGPT) and total bilirubin <3 × upper limit of normal
* The patient and/or their parent/legal guardian is willing and able to provide signed informed consent
* Patients who are sexually active must be willing to abstain from sexual intercourse or agree to use an approved form of contraception while receiving plerixafor and/or standard mobilization treatment and for at least 3 months following any plerixafor treatment

Exclusion Criteria:

* Any form of leukemia
* A co-morbid condition which, in the view of the Investigator, renders the patient at high-risk from treatment complications
* Previous stem cell transplantation
* Persistent high percentage marrow involvement prior to mobilization will be prohibited.
* On-going toxicities (excluding alopecia) Grade ≥2 resulting from prior chemotherapy
* Acute infection
* Fever (temperature >38.5°C) - if fever is between 37°C and 38.5°C, infection must be excluded as a cause
* Known HIV seropositivity, AIDS, hepatitis C or active hepatitis B infections
* Positive pregnancy test in post pubertal girls
* History of clinically significant cardiac abnormality or arrhythmia
* Use of an investigational drug which is not approved in any indication either in adults or pediatrics within 2 weeks prior to the first dose of G-CSF to be administered as part of the patient's planned standard mobilization regimen, and/or during the study up until engraftment of the transplant. If patients are on investigational drugs as part of their anti-cancer regimen, this should be discussed with the Sponsor before screening. Drugs approved for other indications that are being used in a manner considered standard of care for this transplant procedure are allowed
* The patient (and/or their parent/legal guardian), in the opinion of the Investigator, is unable to adhere to the requirements of the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2014-03-03; Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving at least a doubling of peripheral blood CD34+ count during Stage 2 | Up to 5 days

SECONDARY OUTCOMES:
Number of days of apheresis required to reach ≥2 × 10^6 CD34+ cells/kg | Up to 5 days
  During Stage 1 and Stage 2
Yield of CD34+ cells for each apheresis | Up to 5 days
  During Stage 1 and Stage 2
Total CD34+ cell yield | Up to 5 days
  During Stage 1 and Stage 2
Percentage of patients proceeding to transplant | Within 6 months of last apheresis
  During Stage 1 and Stage 2
Percentage of patients successfully engrafting | 3, 6, 12 and 24 months post-transplant
  During Stage 1 and Stage 2
Percentage of patients with durable engraftment | 3, 6, 12 and 24 months post-transplant
  During Stage 1 and Stage 2
Summary of adverse events (AEs) | Up to 24 months after last transplant or 24 months after last dose (for patients that do not transplant within 6 months of last apheresis)
  During Stage 1 and Stage 2
Duration of hospitalizations (planned or unplanned) | Throughout the duration of the study
  During Stage 1 and Stage 2
Mobilization of tumor cells into peripheral blood | Up to 5 days
  During Stage 1 and Stage 2
Relapse rates | 3, 6, 12 and 24 months post-transplant
  During Stage 1 and Stage 2
Occurrence of secondary malignancies | 3, 6, 12 and 24 months post-transplant
  During Stage 1 and Stage 2
Incidence of primary and secondary graft failure | 3, 6, 12 and 24 months post-transplant
  During Stage 1 and Stage 2
Time to secondary graft failure | Up to 24 months post-transplant
  During Stage 1 and Stage 2
Survival rates | 3, 6, 12 and 24 months post-transplant
  During Stage 1 and Stage 2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (27):
- Investigational Site Number 51, Ghent, Belgium
- Czechia (2):
  - Investigational Site Number 81, Brno
  - Investigational Site Number 82, Praha 5 - Motol
- Investigational Site Number 61, København Ø, Denmark
- France (2):
  - Investigational Site Number 42, Lyon
  - Investigational Site Number 43, Paris
- Germany (5):
  - Investigational Site Number 33, Frankfurt am Main
  - Investigational Site Number 34, Freiburg im Breisgau
  - Investigational Site Number 35, Hamburg
  - Investigational Site Number 31, Hanover
  - Investigational Site Number 36, München
- Investigational Site Number 83, Budapest, Hungary
- Israel (2):
  - Investigational Site Number 92, Petah Tikva
  - Investigational Site Number 91, Tel Aviv
- Italy (5):
  - Investigational Site Number 21, Genova
  - Investigational Site Number 24, Milan
  - Investigational Site Number 23, Padua
  - Investigational Site Number 22, Roma
  - Investigational Site Number 26, Torino
- Netherlands (2):
  - Investigational Site Number 72, Amsterdam
  - Investigational Site Number 71, Rotterdam
- Poland (2):
  - Investigational Site Number 85, Krakow
  - Investigational Site Number 84, Wroclaw
- Spain (2):
  - Investigational Site Number 94, Barcelona
  - Investigational Site Number 93, Madrid
- United Kingdom (2):
  - Investigational Site Number 11, Birmingham
  - Investigational Site Number 13, Glasgow

REFERENCES:
- [Derived] Sebastien B, Cheverton P, Magnin C, Aouni J, Castan R. Development and validation of a predictive model to guide the use of plerixafor in pediatric population. Bone Marrow Transplant. 2022 Dec;57(12):1827-1832. doi: 10.1038/s41409-022-01831-2. Epub 2022 Sep 26. PMID 36163427
- [Derived] Morland B, Kepak T, Dallorso S, Sevilla J, Murphy D, Luksch R, Yaniv I, Bader P, Rossler J, Bisogno G, Maecker-Kolhoff B, Lang P, Zwaan CM, Sumerauer D, Krivan G, Bernard J, Liu Q, Doyle E, Locatelli F. Plerixafor combined with standard regimens for hematopoietic stem cell mobilization in pediatric patients with solid tumors eligible for autologous transplants: two-arm phase I/II study (MOZAIC). Bone Marrow Transplant. 2020 Sep;55(9):1744-1753. doi: 10.1038/s41409-020-0836-2. Epub 2020 Mar 3. PMID 32127657